CLINICAL TRIAL: NCT04226430
Title: Effect of a Novel Extracorporeal Cytokine Apheresis Method on Endocan, Copeptin and Interleukin-6 Levels in Sepsis: an Observational Prospective Study.
Brief Title: Effect of Cytosorb on Blood Levels of Inflammatory Biomarkers of Sepsis.
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Berna Kaya Ugur, Assistan Professor, University of Gaziantep
Other Study IDs: TF.18.43
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Sepsis; Cytokine Storm
Keywords: Endocan; Copeptin; Interleukin-6; Cytosorb; Sepsis
MeSH Terms: conditions — Sepsis; Cytokine Release Syndrome; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Sera obtained from arterial blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Before cytosorb: Arterial blood samples were taken from patients before the Cytosorb therapy course.
  Interventions: Device: Cytokine aphaeresis
- after cytosorb: Arterial blood samples were taken from patients immediately after the Cytosorb therapy course.
  Interventions: Device: Cytokine aphaeresis

INTERVENTIONS:
Device: Cytokine aphaeresis — The Cytosorb cartridge was either used alone in hemoperfusion mode or, if renal replacement therapy was clinically indicated, inserted proximally into a conventional continuous veno-venous hemofiltration (CVVH) or continuous veno-venous hemodiafiltration (CVVHDF) circuit. Before the start of the Cytosorb therapy, adequate anti-coagulation was confirmed when target partial thromboplastin time (PTT) of 60±80 seconds, or an activated clotting time (ACT) of 180±210 seconds was achieved with systemic heparin. Antibiotics were administered after each Cytosorb therapy whenever possible.
  Other Names: Cytosorb

SUMMARY:
Background: There is still an evident need for useful biomarkers and effective therapeutic approaches regarding the challenging management of sepsis. The aim of the study is to evaluate the effect of each Cytosorb hemoadsorption therapy course on blood levels of inflammatory biomarkers of sepsis including endocan, copeptin, interleukin-6, procalcitonin, C-reactive protein.

DETAILED DESCRIPTION:
This observational prospective study included patients, who were diagnosed with sepsis and treated in the reanimation ICU of Gaziantep University Hospital with Cytosorb therapy between June 1st, 2016 and June 30th, 2017. Sepsis was diagnosed according to The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3).

Exclusion criteria of the study were: (i) cardiovascular disease, (ii) multiple traumas, (iii) malignancies, (v) incomplete clinical data.

Approval of the ethical committee (ethical committee approval number 2018/04-02) was obtained. Written informed consent was taken from each patient or their next-of-kin. Patient demographics including age, gender, and origin of sepsis were recorded. Arterial blood samples were taken from patients before and immediately after the Cytosorb therapy course.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who were diagnosed with sepsis and treated in the reanimation ICU of Gaziantep University Hospital with Cytosorb therapy (Sepsis was diagnosed according to The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3))

Exclusion Criteria:

* cardiovascular disease,
* multiple traumas
* malignancies
* incomplete clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This observational prospective study included patients, who were diagnosed with sepsis and treated in the reanimation ICU of Gaziantep University Hospital.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Effect of a novel extracorporeal cytokine apheresis method on endocan levels in sepsis | 13 months
  The effect of each Cytosorb hemoadsorption therapy course on blood levels of endocan, an inflammatory biomarker of sepsis.
Effect of a novel extracorporeal cytokine apheresis method on copeptin levels in sepsis | 13 months
  The effect of each Cytosorb hemoadsorption therapy course on blood levels of copeptin, an inflammatory biomarker of sepsis.
Effect of a novel extracorporeal cytokine apheresis method on interleukin-6 levels in sepsis | 13 months
  The effect of each Cytosorb hemoadsorption therapy course on blood levels of interleukin-6, an inflammatory biomarker of sepsis.

IPD SHARING:
Plan to Share IPD: No
All data included in the manuscript that will be published.